CLINICAL TRIAL: NCT04885894
Title: An Examination of Cognitive Fatigue Using Functional Neuroimaging
Status: Recruiting | Type: Observational
Sponsor: Kessler Foundation (Other)
Collaborators: Celgene (Industry); Hackensack Meridian Health (Other); St. Barnabas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: R-1150-21
Record Dates: First submitted 2021-05-11; First posted 2021-05-13 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ozanimod

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MS Zeposia: Individuals with MS who will begin taking Zeposia as part of standard care.
  Interventions: Drug: Zeposia
- MS High dose efficacy medication: Individuals with MS who will begin taking high dose efficacy oral medication as part of standard of care.
- Healthy Control: Healthy controls, all of whom will be matched on age, education and gender to the MS groups.

INTERVENTIONS:
Drug: Zeposia — Participants with MS will be divided into two treatment groups: those who will begin to take Zeposia, and those who plan to be begin treatment with high dose oral efficacy medication. The HC group will be free of neurological disease or injury and will be matched to the MS groups for age, gender, and education.
  Groups: MS Zeposia

SUMMARY:
The purpose of this research study is to investigate the effectiveness of MS Disease modifying medications on cognitive fatigue in persons with relapsing remitting multiple sclerosis (RRMS). Cognitive fatigue is the kind of fatigue that occurs after intense mental concentration as after a session of problem solving.

DETAILED DESCRIPTION:
The researchers aim is to investigate the effects of disease modifying treatments on cognitive fatigue and on specific brain areas that have been shown to underlie cognitive fatigue in individuals with Multiple Sclerosis (MS). The researchers will investigate the effects on the cognitive fatigue that develops during the performance of a demanding task, and also on how cognitive fatigue changes as a function of duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-64.
* Relapsing remitting multiple sclerosis
* Been newly prescribed a new disease modifying medication for MS (either Zeposia or other high dose oral efficacy medication)
* or healthy volunteer who can speak English fluently.

Exclusion Criteria:

* History of head injury, stroke, seizures, or any other significant neurological event other than MS
* Flare up of MS symptoms within the past month.
* History of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder.
* Pacemaker or other implanted electrical device, brain stimulator, aneurysm clip (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and internal hearing aids [cochlear implants]), permanent eyeliner, implanted delivery pumps, or shrapnel fragments.
* left handed.
* Not able to have an MRI

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with Relapsing Remitting Multiple Sclerosis and Healthy Controls
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Brain activation (BOLD signal) | Measured for change at 3 time points (before, six months and 12 months after intervention)
  A change in brain activation as measured with functional magnetic resonance imaging through blood oxygen level dependent signal will be measured in association with cognitive fatigue (as measured by the Visual Analogue scale during performance of the modified Symbol Digit Modality and Modified Fatigue Impact Scale).

SECONDARY OUTCOMES:
Fatigue Onset | Measured for change at 3 time points (before, six months and 12 months after intervention)
  A change in the speed with which modified Symbol Digit Modality task (a cognitively demanding task) induces fatigue in MS (as measured by the Visual Analogue scale and Modified Fatigue Impact Scale).

CONTACTS AND LOCATIONS:
Overall Officials: John DeLuca, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No